CLINICAL TRIAL: NCT00150644
Title: A Phase 2, 12-Week, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Effects of J867 on Uterine Artery Blood Flow and the Morphology of the Endometrium, Myometrium, and Uterine Leiomyomata in Subjects With Uterine Leiomyomata Scheduled for Hysterectomy.
Brief Title: A Study to Evaluate the Effects of Asoprisnil(J867) in Women With Uterine Fibroids Who Are Scheduled for a Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C02-003
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Uterine Fibroids; Leiomyoma
Keywords: Fibroid Uterus; Leiomyoma; Uterine Fibroids; Hysterectomy; Asoprisnil
MeSH Terms: conditions — Leiomyoma | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asoprisnil — Asoprisnil 10mg Tablet, oral Daily for 12 weeks
  Other Names: J867
  Arms: 1
Drug: Asoprisnil — Asoprisnil 25 mg Tablet, oral Daily for 12 weeks
  Other Names: J867
  Arms: 2
Drug: Placebo — Placebo Tablet, oral Daily for 12 weeks
  Arms: 3

SUMMARY:
The objective of this study is to evaluate the effects of 10 mg and 25 mg doses of asoprisnil, compared to placebo, taken daily for 12 weeks, on uterine blood flow and the morphology of the endometrium and uterine fibroids.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of uterine fibroids. The objective of this study is to determine the effects of asoprisnil in uterine fibroid growth suppression. Full thickness biopsies obtained from surgical procedures will allow the assessment of asoprisnil's effects on the basalis, the myometrium, and on endometrial angiogenesis. Various other exploratory immunohistological and biochemical specimens will be collected to evaluate the mechanisms of action of asoprisnil in the endometrium, the myometrium, and in uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, at least 18 years of age
* Diagnosis of uterine fibroid(s), confirmed by ultrasound
* History of menstrual cycles between 17 and 42 days
* Otherwise in good health
* Scheduled for a hysterectomy at the end of the treatment period
* Negative pregnancy test
* Agrees to double barrier method of contraception
* Pap test with no evidence of malignancy or pre-malignant changes
* Endometrial biopsy with no significant histological disorder

Exclusion Criteria:

* Less than 3 months after having a baby or breast-feeding
* Any abnormal lab or procedure result the study-doctor considers important
* Severe reaction(s) to or are currently using any hormone therapy
* History of cancer or alcohol or drug abuse
* Diagnosis of Polycystic Ovary Syndrome
* History of prolactinoma
* Current use of Intrauterine Device
* Significant gynecological disorder
* Uterine size > 32 weeks gestation
* Current diagnosis of endometriosis
* Uterine artery embolization within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-07; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the Final Visit in uterine artery blood flow as determined by change in Resistance Index. | Final visit

SECONDARY OUTCOMES:
Change from baseline in uterine artery blood flow as determined by change in Pulsatility Index. | Final Visit
Morphological changes in the endometrium, myometrium and uterine fibroids. | Final Visit
Change from baseline in menstrual pictogram score. | Final Month
Percent change from baseline in volume of the largest fibroid. | Final Visit
Endometrial thickness (post-treatment histologic evaluation). | Final Visit
Change from baseline in endometrial thickness by transvaginal ultrasound. | Final Visit
Percent of ovulatory subjects. | Final Month
Change from baseline in the Uterine Fibroid Symptom-Quality of Life total symptom severity score and the Uterine Fibroid Symptom-Quality of Life total score. | Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott

REFERENCES:
- [Result] Williams AR, Critchley HO, Osei J, Ingamells S, Cameron IT, Han C, Chwalisz K. The effects of the selective progesterone receptor modulator asoprisnil on the morphology of uterine tissues after 3 months treatment in patients with symptomatic uterine leiomyomata. Hum Reprod. 2007 Jun;22(6):1696-704. doi: 10.1093/humrep/dem026. Epub 2007 Mar 5. PMID 17339234